CLINICAL TRIAL: NCT04282681
Title: XLTCS - Accelerometer Data Collection in an Epilepsy Monitoring Unit (EMU)
Acronym: XLTCS
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor decision due to clinical strategy changes
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Other Study IDs: LNE-800
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Epilepsy, Tonic-Clonic
MeSH Terms: conditions — Epilepsy, Tonic-Clonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Accelerometer Live-Streaming Tool — The only 'intervention' that will take place is the placement of the XLS tool(s) on the upper left chest and/or left wrist of the patient.

SUMMARY:
The primary objective of this study is to collect accelerometer data from subjects monitored in an EMU with concurrent video EEG.

DETAILED DESCRIPTION:
XLTCS (LNE-800) is an international multicenter prospective data collection study to gather accelerometer data. The population under the study comprises patients monitored in an Epilepsy Monitoring Unit (EMU) with concurrent video EEG and who are expected to have at least one seizure with tonic-clonic convulsive movement.

A maximum of one hundred and fifty (150) patients will be enrolled and will wear an accelerometer, and up to 6 sites may participate in this study. The total enrollment period will take approximately 2 years.

Once the accelerometer was adhered to the subject, subjects will be followed for a minimum of 2 days and a maximum of 10 days.

Subject participation will run concurrently with the EMU admission. Exit from the study occurs when the subject's stay in the EMU is completed or the subject is withdrawn or withdraws from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Four (4) years of age or older.
2. Admitted to an Epilepsy Monitoring Unit for video EEG monitoring.
3. Based on medical history, expected to have at least one seizure with tonic-clonic convulsive movement during the EMU stay as determined by the investigator.
4. Capable of understanding and willing to comply with instructions and study procedures.
5. Subject or guardian must be willing and able to complete informed consent/assent.

Exclusion Criteria:

1. Based on medical history, expected to have only non-epileptic events during the EMU stay as determined by the investigator.
2. Based on medical history, known to have only absence seizures.
3. Medical or psychiatric condition that in the investigator's judgment would prevent the subject's successful completion of the study.
4. Participants with known hypersensitivity or skin sensitivity conditions that will preclude attachment of the accelerometer.
5. Participants who are also taking part in another clinical trial that could confound the results of the study; these patients can be included into the study only if LivaNova has provided written approval.

Ages: 4 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have been admitted to an EMU for video EEG monitoring (independent of this study) who are expected to have at least one seizure with tonic-clonic convulsive movement.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-16 (Estimated); Primary Completion 2021-08-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate accelerometer data and tonic-clonic seizure data | 1.5 years
  The study will evaluate accelerometer data and tonic-clonic seizure data that was collected during the patients' EMU admission. The sample size is not based on a statistical power calculation, thus no primary endpoint is defined in the clinical investigation plan.

CONTACTS AND LOCATIONS:
Overall Officials: Krisl Vonck, Principal Investigator — University Hospital, Ghent
Locations (1):
- Universitair Ziekenhuis Gent, Ghent, Belgium